CLINICAL TRIAL: NCT05542264
Title: A Double-Blind, Randomized, Multiple Dose Study of Weight Associated Parameters: SEP-363856 vs Prior Antipsychotic (PA) Standard of Care in Subjects With Schizophrenia Suffering From Metabolic Dysregulation
Brief Title: A Clinical Study That Will Assess the Effect of SEP-363856 or Prior Antipsychotic (PA) Standard of Care on Body-weight Associated Parameters in Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-122
Record Dates: First submitted 2022-08-15; First posted 2022-09-15 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856; Risperidone; Olanzapine; Quetiapine Fumarate; Aripiprazole

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Multiple Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole) (Active Comparator)
  Interventions: Drug: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole)
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 will be supplied as over-encapsulated tablets. Multiple tablets may be required to achieve a single dose.
  Arms: SEP-363856
Drug: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole) — PA will be prepared by the pharmacy staff according to the patient's prescribed treatment and will be orally administered. Multiple tablets or capsules may be required to achieve a single dose.
  Arms: Prior antipsychotic (risperidone, olanzapine, quetiapine or aripiprazole)

SUMMARY:
A Clinical Study that will look at an investigational medication, SEP-363856 (called "study medication") in patients with schizophrenia, and assess wether it affectsbody-weight associated parameters. This study is accepting male and female participants age 18 years to 65 years. This study will be conducted in approximately 6 study sites in the United States. Participation could last up to 13 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, multiple dose study in male and female adult subjects with schizophrenia. Subjects will undergo structural magnetic resonance abdominal imaging (MRI) scans as well as hyperinsulinemic euglycemic clamp (HEC) also known as "glucose clamp", after the check-in and towards the end of the treatment phase. Subjects will be randomized to SEP-363856 or their prior antipsychotic (PA). Subjects randomized to SEP-363856 will undergo blinded wash out of their PA, subsequent SEP-363856 blinded titration and 15 day of well tolerated SEP-363856 exposure. Subjects randomized to their prior antipsychotic (PA), will undergo pseudo PA washout, followed by pseudo-titration and 15 day of well tolerated PA exposure. Subjects will be discharged after subject is stable. All subjects will return to the clinic 7 + 2 days post discharge for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria: This is not an all inclusive list

* Male or female subjects between 18 and 65 years of age, inclusive at time of consent.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of schizophrenia as established by clinical interview, using the DSM-5 as a reference and confirmed using the Structured Clinical Interview for DSM-5, Clinical Trials Version [SCID-CT]).
* Subject must have a Positive and negative symptoms scale (PANSS) total score ≤ 80 at Screening and a score of ≤ 4 on the following PANSS items at Screening: P7 (hostility) and G8 (uncooperativeness)
* Subject must have a Clinical Global Impressions - Severity (CGI-S) score ≤ 4 (normal to moderately ill) at Screening.
* Subject must be receiving risperidone, olanzapine, quetiapine or aripiprazole as treatment for schizophrenia at the time of Screening.

Exclusion Criteria: This is not an all inclusive list

* Subject has a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia or intellectual disability (IQ < 70).
* Subject has attempted suicide within 12 months prior to Screening.
* Subject answers "yes" to "Suicidal Ideation" Items 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS at Screening (ie. in the past 1 month) or at any subsequent C-SSRS assessment prior to dosing (ie, since last visit).
* Subject is at risk of harming him/herself or others according to the Investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Insulin stimulated change in glucose disposal rate during the steady state of the low dose hyperinsulinemic euglycemic clamp (HEC), baseline to end of the treatment | up to 8 weeks
Insulin stimulated change in glucose disposal rate during the steady state of the high dose hyperinsulinemic euglycemic clamp (HEC) baseline to end of the treatment. | up to 8 weeks
Change in liver proton density fat fraction (PDFF), baseline to end of the treatment | up to 8 weeks
Change in fat content in muscles of interest, baseline to end of the treatment | up to 8 weeks
Change in Liver Fibroinflammation, baseline to end of the treatment | up to 8 weeks
Change in Liver Volume from baseline to end of treatment | up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Woodland International Research Group, Little Rock, Arkansas
  - Shari DeSilva, Rogers, Arkansas
  - Midwest Clinical Research Center, Dayton, Ohio
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com